CLINICAL TRIAL: NCT00006077
Title: Effects of Monoamine Reuptake Inhibitor NS2330 in Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000187; 00-N-0187
Record Dates: First submitted 2000-08-04; First posted 2000-08-07 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-07

CONDITIONS: Parkinson's Disease
Keywords: Clinical Trial; Dyskinesias; Levodopa Infusion; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — Levodopa; Domperidone

INTERVENTIONS:
Drug: NS2330
Drug: Levodopa and Domperidone

SUMMARY:
This study will evaluate the effects of an experimental drug called NS2330 on Parkinson's disease symptoms and on dyskinesias (involuntary movements) that develop as a result of long-term treatment with levodopa. This drug prevents the neurotransmitter dopamine from entering nerve cells.

Patients between 18 and 75 years old who have moderately advanced Parkinson's disease and motor problems resulting from levodopa therapy may be eligible for this 5-week study. Candidates will have a complete medical history and physical examination with a detailed neurological evaluation. If needed, some patients will undergo a magnetic resonance imaging (MRI) or computerized tomography (CT) scan of the brain and a chest X-ray. All patients will have blood and urine tests and an electrocardiogram (EKG) and will take a written test for evaluation of depression.

Patients enrolled in the study will, if possible, stop taking all antiparkinson medications except levodopa (Sinemet) for one month before the study begins and through its duration. For the first 1 to 3 days, patients will undergo a levodopa "dose-finding" procedure. For this study, patients will stop taking their usual oral levodopa medicine and instead will have levodopa infused through a vein for up to 12 hours. During the infusions, the drug dose will be increased slowly until either 1) parkinsonism symptoms improve, 2) dyskinesias appear, 3) unacceptable side effects occur, or 4) the maximum study dose is reached.

When the patient's optimal dose is determined, treatment will begin. Patients will take three pills containing NS2330 or placebo (a look-alike pill with no active ingredient) 3 days a week for up to 5 weeks, in addition to their regular levodopa medication. All participants will receive placebo at some point in the study; some patients will receive only placebo throughout the entire 5 weeks.

On treatment days, patients will have a brief medical examination before receiving the drug and will then be monitored for side effects for about 6 to 8 hours after taking the drug. At the beginning of weeks 2 and 5, the levodopa infusions will be repeated at the previously determined optimum rate. Throughout the study, parkinsonism symptoms, dyskinesias and depression will be evaluated. Blood and urine samples will be collected each week for standard safety tests, and blood will also be drawn periodically to measure NS2330 levels.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the acute effects of a potent inhibitor of dopamine reuptake on the severity of parkinsonian signs and levodopa-associated motor response complications in patients with Parkinson's disease. In a controlled proof-of-principle clinical trial, the efficacy of NS2330 will be assessed through the use of validated motor function scales. Safety will be monitored by means of frequent clinical evaluations and laboratory tests.

ELIGIBILITY:
INCLUSION CRITERIA

Male and Females are eligible for this study.

Ages 18-75.

Women must be at least one year post-menopausal or using an adequate contraceptive method for at least one month prior to and during participation in the study.

All will carry the diagnosis of idiopathic Parkinson's disease based on the presence of a characteristic clinical history and neurologic findings.

All will have relatively advanced disease with levodopa-associated motor response complications, including wearing-off fluctuations and peak-dose dyskinesias.

EXCLUSION CRITERIA

The presence or history of any medical condition that can reasonably be expected to subject the patient to unwarranted risk.

Any clinically significant laboratory abnormalities including liver enzyme elevations more than twice the upper limit of normal, or neutropenia (wbc less than 4000).

Patients with diphasic or end-of dose dyskinesias or disabling dystonia.

Patients who are unable to be treated with levodopa/carbidopa alone or a single, relatively short-acting dopamine agonist.

Patients with any form of Parkinsonism other than idiopathic PD or with a diagnosis of dementia or major psychiatric disorder. Individuals with mild to moderate depression will be sought for this study, unless their depressive disorder currently requires regular medical therapy.

Patients who are on unacceptable prior/concomitant medications.

Pregnant women

Those who are not practicing effective birth control.

Patients with prior bilateral neurosurgical intervention for the treatment of Parkinsonian symptoms, i.e. deep brain stimulation, pallidotomy, fetal tissue transplantation as well as patients at risk for symptomatic hypotension, cardiac arrhythmia, and/or myocardial ischemia secondary to intravenous levodopa challenge or NS2330 therapy.

Patients who have taken an investigational drug within the last two months prior to randomization.

Previous participation in any NS 2330 study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2000-08; Study Completion 2003-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bernheimer H, Birkmayer W, Hornykiewicz O, Jellinger K, Seitelberger F. Brain dopamine and the syndromes of Parkinson and Huntington. Clinical, morphological and neurochemical correlations. J Neurol Sci. 1973 Dec;20(4):415-55. doi: 10.1016/0022-510x(73)90175-5. No abstract available. PMID 4272516
- [Background] Mizuno Y, Mori H, Kondo T. Parkinson's disease: from etiology to treatment. Intern Med. 1995 Nov;34(11):1045-54. doi: 10.2169/internalmedicine.34.1045. PMID 8774962
- [Background] Chase TN, Oh JD, Blanchet PJ. Neostriatal mechanisms in Parkinson's disease. Neurology. 1998 Aug;51(2 Suppl 2):S30-5. doi: 10.1212/wnl.51.2_suppl_2.s30. PMID 9711978